CLINICAL TRIAL: NCT05589441
Title: Nebulized Salbutamol Facilitate Management of Hyperkalemia Postreperfusion During Liver Transplantation: a Single-center, Randomized, Positive-controlled Clinical Study
Brief Title: Nebulized Salbutamol Facilitate Management of Hyperkalemia Postreperfusion During Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2019-021
Record Dates: First submitted 2022-09-18; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-09

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Albuterol; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulized inhalation of salbutamol group (Experimental): 10 mg salbutamol diluted to 2 ml with distilled water and inhaled as aerosolized for 15 min before the start of the hepatic-free phase.
  Interventions: Drug: salbutamol
- Insulin complex glucose group (Experimental): Intravenous injection of 8U of insulin complex 10% glucose solution 250 ml before the start of the hepatic phase was completed in 15 minutes.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: salbutamol — 10 mg salbutamol diluted to 2 ml with distilled water and inhaled as aerosolized for 15 min before the start of the hepatic-free phase.
  Other Names: Nebulized inhalation of salbutamol
  Arms: Nebulized inhalation of salbutamol group
Drug: Insulin — Intravenous injection of 8U of insulin complex 10% glucose solution 250 ml before the start of the hepatic phase was completed in 15 minutes.
  Other Names: Insulin complex glucose group
  Arms: Insulin complex glucose group

SUMMARY:
The therapeutic effect of nebulized salbutamol on hyperkalemia during reperfusion in liver transplantation patients. Secondary research objectives: To observe the results of blood gas analysis, changes in urinary potassium and hemodynamic parameters, and the incidence of reperfusion syndrome in liver transplantation, and to observe the incidence of postoperative pulmonary complications during the 7-day follow-up. To explore the effect of aerosol inhalation of salbutamol on new liver reperfusion syndrome in patients with liver transplantation, and to provide a theoretical basis for clinical treatment.

DETAILED DESCRIPTION:
1. Research background 1.1 Study disease Hyperkalemia during reperfusion in patients with end-stage liver disease undergoing liver transplantation 1.2 Research status at home and abroad 1.2.1 Hyperkalemia in the perioperative period of liver transplantation and hyperkalemia caused by DCD donor liver Hyperkalemia refers to a state in which the concentration of potassium ions in the patient;s serum exceeds 5 mmol/L.Clinical symptoms include muscle twitches, spasms, weakness, ascending paralysis, ECG changes, and heart rhythm.

   Severe hyperkalemia can be life-threatening in the form of abnormalities. Hyperkalemia is a common complication in orthotopic liver transplantation. Immediate blood potassium in new liver reperfusion can be as high as 7 mmol/L to 8 mmol/L. Especially in patients with renal insufficiency, the clinical manifestations are more dangerous, which can lead to serious complications. Arrhythmias and even cardiac arrest. There are several reasons for the occurrence of hyperkalemia during liver transplantation: 1. Severe metabolic acidosis in the anhepatic phase, resulting in increased H+-K+ exchange on the cell membrane; 2. Poor coagulation function in patients undergoing liver transplantation, Intraoperative red blood cell transfusion volume is large, resulting in the increase of exogenous potassium ions; 3 UW organ protection solution for liver transplantation contains a large amount of potassium ions, which enter the blood circulation after reperfusion, resulting in post-reperfusion hyperkalemia . Since January 1, 2015, organ donation after the death of a citizen (DCD) has become the only legal source of organ transplant donors in China. Recent studies have shown that DCD donors are the main source of hyperkalemia after liver transplant reperfusion. This is an independent risk factor for liver disease, which is due to the long warm ischemia time in the liver of DCD donors, and the hypoxic injury of hepatocytes is more serious, and the damage of oxygen free radicals after reperfusion will cause potassium ions to be released from hepatocytes. Under this circumstance, it is particularly important to prevent and treat hyperkalemia after reperfusion to ensure the safety of perioperative anesthesia in patients with liver transplantation.

   1.2.2 Treatment of hyperkalemia At present, the methods of treating hyperkalemia routinely used in clinic are as follows: 1 Membrane stabilizer Commonly used are calcium gluconate and calcium chloride. Hyperkalemia increases the action potential threshold of cardiomyocytes and causes myocardial membrane instability. Calcium ions can counteract this situation by restoring the transmembrane voltage gradient of cardiomyocytes and reduce the toxicity of cardiomyocytes caused by hyperkalemia. 2 To promote the excretion of potassium ions The most commonly used are the use of diuretics, hemodialysis, potassium-lowering resin. 3 Redistribution of potassium ions in and out of cells Insulin combined with glucose infusion, nebulized inhalation or intravenous salbutamol. However, not every method is suitable for liver transplantation. Intravenous calcium injection can stabilize the cell membrane against the toxic effect of high potassium on the myocardium, but it cannot reduce the serum potassium ion concentration, and there is a risk of bradycardia. Side effects: Most patients with end-stage liver disease have hepatorenal syndrome, and the effect of diuretics is limited, and after extensive use, it will aggravate the occurrence of cellular metabolic acidosis, and even increase serum potassium. Hemodialysis is one of the most effective treatments for hyperkalemia, but its use is limited in liver transplantation, and a dialysis pipeline needs to be established in advance, and the use of heparin during dialysis to prevent thrombosis in the pipeline will affect the coagulation function of patients and cause intraoperative complications. Bleeding increases and is less used in liver transplantation; potassium-lowering resin has a slow onset and limited effect, and needs to be taken from the gastrointestinal tract and cannot be used in liver transplantation; patients with end-stage liver disease usually have insulin resistance;, Intravenous infusion of insulin compounded with glucose, the dose of administration is difficult to control, the therapeutic effect is unreliable, and it is easy to cause severe fluctuations in the blood glucose level of patients during the perioperative period. Studies have found that salbutamol can transport potassium ions in serum to liver cells and skeletal muscle cells by activating sodium-potassium-ATPase and NKCC1 Na+-K+-2Cl- co-transporter, thereby reducing serum potassium ion concentration.

   1.2.3 The application prospect of nebulized salbutamol in the perioperative period of liver transplantation Salbutamol is an adrenergic β-receptor agonist, because it can selectively stimulate the β2-receptor of bronchial smooth muscle, it is a strong bronchodilator, and it is mainly used in the clinical prevention and treatment of bronchial asthma or asthmatic bronchitis , improve the patient ventilation function. Recent studies found that salbutamol can transport potassium ions in serum to liver cells and skeletal muscle cells by activating sodium-potassium-ATPase and NKCC1 Na+-K+-2Cl- co-transporters, reducing serum potassium ions. concentration. Among them, there are two kinds of administration modes of salbutamol: intravenous injection and atomization inhalation, among which the method of atomization inhalation has good effect and small side effects. In patients with end-stage renal disease and hyperkalemia, the serum potassium ion concentration decreased by 0.6 mmol/L 30 minutes after inhalation of 10 mg of salbutamol, and decreased by 1 mmol/L one hour later. However, there is no report on its application in the treatment of hyperkalemia during reperfusion of liver transplantation. All liver transplantation operations are performed under general anesthesia with endotracheal intubation. It is small, convenient and easy to operate, and intraoperative atomized inhalation of salbutamol can also stimulate β receptors, increase heart rate, and resist the occurrence of reperfusion syndrome, which has good research opportunities and clinical application value.

   1.3 Preliminary research results of the project team

   The investigators liver transplantation anesthesia team has now conducted a preliminary experiment in 10 cases of liver transplantation by inhalation of salbutamol before the anhepatic phase. The concentration of serum potassium can be significantly reduced 30 minutes after inhalation. The data are as follows:

   Items 5min before inhalation(Blood potassium:4.35±0.26mmol/L 5min after inhalation(Blood potassium:4.34±0.30mmol/L 10min after inhalation(Blood potassium:4.15±0.33mmol/L 15min after inhalation(Blood potassium:4.05±0.29mmol/L 30min after inhalation(Blood potassium:3.6±0.31**mmol/L 45min after inhalation(Blood potassium:3.25±0.41**mmol/L 30s after reperfusion(Blood potassium:5.21±0.68mmol/L 5 min after reperfusion(Blood potassium:3.91±0.55mmol/L 30min after reperfusion(Blood potassium:3.53±0.49mmol/L (mmol/L)
2. Research objectives 2.1 Main research objectives To observe the effect of nebulized inhalation of salbutamol in the treatment of hyperkalemia during liver transplantation and reperfusion 2.2 Secondary research objectives and exploratory research objectives The changes in blood gas, urine potassium and hemodynamic parameters during surgery in liver transplant patients were observed, and the incidence of postoperative complications was observed 7 days after surgery. To explore the effect of nebulized inhalation of salbutamol on liver transplant patients on intraoperative reperfusion syndrome and postoperative lung complications, and to provide a theoretical basis for clinical treatment.
3. Research Overview 3.1 Study Type Randomized, double-blind, parallel controlled clinical trial Single-centered, prospective, randomized, controlled studies Single Center: The First Affiliated Hospital of Jiaotong University Random: Generate a random grouping table by a random program. Make sealed envelopes with random information based on random grouping tables. Pay attention to age, sex, ASA grade, and surgeon balance at random. After the patient is selected and randomized, open the envelope according to the corresponding random number to obtain the random number.

Positive controls: nebulized inhalation of salbutamol group and insulin complex glucose group in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 70 years old;
* Cardiac function grades I to III (NYHA standard);
* Plan to undergo orthotopic liver transplantation;
* Serum potassium ion concentration greater than 4 mmol/h at the beginning of anhepatic phase;
* Those who are willing to sign the informed consent form.

Exclusion Criteria:

* Intraoperative CRRT patients;
* Those who are allergic to the test drug;
* refuse to join the trial investigator;
* Patients who are participating in other clinical trials, the researchers believe that other reasons are not suitable for clinical trials.
* Anyone with any of the above conditions cannot be selected for this trial.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-28 (Estimated); Primary Completion 2023-10-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Blood potassium concentration,mmol/L | measured blood gas at 5 minutes before treatment
  Patients who met the inclusion and exclusion criteria were enrolled and assigned random numbers. After randomization, the intervention was given at the beginning of the anhepatic phase according to the grouping
Blood potassium concentration,mmol/L | measured blood gas at 5 minutes after treatment
  Patients who met the inclusion and exclusion criteria were enrolled and assigned random numbers. After randomization, the intervention was given at the beginning of the anhepatic phase according to the grouping
Blood potassium concentration,mmol/L | measured blood gas at 10 minutes after treatment
  Patients who met the inclusion and exclusion criteria were enrolled and assigned random numbers. After randomization, the intervention was given at the beginning of the anhepatic phase according to the grouping
Blood potassium concentration,mmol/L | measured blood gas at 15 minutes after treatment
  Patients who met the inclusion and exclusion criteria were enrolled and assigned random numbers. After randomization, the intervention was given at the beginning of the anhepatic phase according to the grouping
Blood potassium concentration,mmol/L | measured blood gas at 30 minutes after treatment
  Patients who met the inclusion and exclusion criteria were enrolled and assigned random numbers. After randomization, the intervention was given at the beginning of the anhepatic phase according to the grouping
Blood potassium concentration,mmol/L | measured blood gas at 45 minutes after treatment
  Patients who met the inclusion and exclusion criteria were enrolled and assigned random numbers. After randomization, the intervention was given at the beginning of the anhepatic phase according to the grouping
Blood potassium concentration,mmol/L | measured blood gas at 60 minutes after treatment
  Patients who met the inclusion and exclusion criteria were enrolled and assigned random numbers. After randomization, the intervention was given at the beginning of the anhepatic phase according to the grouping
Blood potassium concentration,mmol/L | measured blood gas at 30 seconds after reperfusion
  Patients who met the inclusion and exclusion criteria were enrolled and assigned random numbers. After randomization, the intervention was given at the beginning of the anhepatic phase according to the grouping
Blood potassium concentration,mmol/L | measured blood gas at 5 minutes after reperfusion
  Patients who met the inclusion and exclusion criteria were enrolled and assigned random numbers. After randomization, the intervention was given at the beginning of the anhepatic phase according to the grouping
Blood potassium concentration,mmol/L | measured blood gas at 30 minutes after reperfusion
  Patients who met the inclusion and exclusion criteria were enrolled and assigned random numbers. After randomization, the intervention was given at the beginning of the anhepatic phase according to the grouping

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wen, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No
Clinical Study Data and Results

REFERENCES:
- [Derived] Ding Y, Wen J, Xiao Y. Comparison of nebulized salbutamol and glucose-insulin for preventing acute hyperkalemia in liver transplantation: a randomized, double-blind trial. J Anesth. 2026 Jan 21. doi: 10.1007/s00540-025-03643-2. Online ahead of print. PMID 41565838